CLINICAL TRIAL: NCT06111911
Title: Detection of High-Risk Human Papilloma Virus in Urine and Cervical Swab Specimens; Comparison Between HPV Diagnostic Kit (Bio Farma) and COBAS 6800 HPV (Roche Molecular Systems)
Brief Title: Detection of High-Risk HPV in Urine and Cervical Swab Specimen Using HPV Diagnostic Kit (Bio Farma)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Protokol-BIO-HPV14-BIOFARMA
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Human Papilloma Virus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urine Specimen (Experimental)
  Interventions: Diagnostic Test: HPV Diagnostic Kit (Bio Farma)
- Cervical Swab Specimen (Experimental)
  Interventions: Diagnostic Test: HPV Diagnostic Kit (Bio Farma)

INTERVENTIONS:
Diagnostic Test: HPV Diagnostic Kit (Bio Farma) — Urine samples (30 ml): collected from each subjects using urine pot. Cervical swab: collected from each subject using cyto brush and stored in special container which preservatives fluid.
  Other Names: COBAS 6800 HPV from Roche Molecular Systems

SUMMARY:
This study is a cross-sectional study to evaluate accuracy of high-risk DNA-HPV testing using HPV Diagnostic Kit (Bio Farma) compared to Standard Kit (COBAS® 6800 HPV from Roche Molecular Systems) RT-PCR based in urine and cervical swab specimens.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active female aged 20-50 years
* Willing to participate in study and signed the informed consent form.

Exclusion Criteria:

* Pregnant women
* History of HIV infection
* On menstruation period
* History of complete HPV vaccination

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
Performance of HPV Diagnostic Kit (Bio Farma) using urine and cervical swab sample | 0 days
  Sensitivity and Specificity of HPV Diagnostic Kita (Bio Farma)

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No